CLINICAL TRIAL: NCT01356524
Title: Relationship Between Mid-luteal Serum Progesterone Levels to Pregnancy Rates in Assisted Reproductive Techniques (ART)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Nardin Aslih MD, Hillel Yaffe Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HYH-28-11
Record Dates: First submitted 2011-05-18; First posted 2011-05-19 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2011-05

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Supplementary progesterone (Active Comparator): Women with mid-luteal progesterone levels that are less than 15 ng/dl will receive higher doses of supplementary progesterone
  Interventions: Drug: Additional vaginal progesterone
- No additional progesterone (No Intervention): No additional progesterone given to women with mid-luteal progesterone levels below 15 ng/dl

INTERVENTIONS:
Drug: Additional vaginal progesterone — The progesterone dose will be raised from 200 mg daily to 300 mg daily
  Arms: Supplementary progesterone

SUMMARY:
In Assisted Reproductive Techniques (ART) there is a need for luteal support using progesterone, estrogen and probably human chorionic gonadotropin (HCG). The optimal route of administration and dose has not yet been determined.

The aim of the study is to investigate whether high levels of mid-luteal serum progesterone are related to higher pregnancy rates in ART cycles. We also plan to investigate whether using higher doses of vaginal progesterone results in higher pregnancy rates.

ELIGIBILITY:
Inclusion Criteria:

* Mid-luteal serum progesterone levels below 15 ng/dl

Exclusion Criteria:

* Does not sign consent form

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2011-07; Primary Completion 2012-07 (Estimated); Study Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
Pregnancy rates | One week

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel